CLINICAL TRIAL: NCT06372418
Title: Enhancing Growth and Development Among Malnourished Infants Recovering From a Serious Illness (IBAMI-2)
Brief Title: Providing Breastfeeding Support After Discharge From Hospital to Improve Growth and Development of Malnourished Infants
Acronym: IBAMI-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KEMRI/SERU/CGMR-C/238/4326
Record Dates: First submitted 2023-07-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Malnutrition, Infant; Breastfeeding, Exclusive
MeSH Terms: conditions — Infant Nutrition Disorders; Breast Feeding | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial:
  Participants will be randomized to either receive Breastfeeding support intervention (BFSI) or standard of care.
Who Masked: Outcomes Assessor
Masking Description: Fieldworkers collecting endpoint data at 6 months of age will be blinded to group allocation to avoid any bias subject to knowledge of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding peer support intervention. (Experimental): In addition to support as currently recommended by the World Health Organization (WHO) and National IMAM guidelines, the intervention arm will receive a homebased individualized face to face support breastfeeding by peer supporters and phone support for 7 weeks post hospital discharge.
  Interventions: Other: Breastfeeding peer support intervention
- Standard of care (Active Comparator): The Control arm will receive post-discharge support as currently recommended by the World Health Organization (WHO) and national IMAM guidelines, including providing linkage to available local breastfeeding support groups.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Breastfeeding peer support intervention — In addition to support as currently recommended by the World Health Organization (WHO) and National IMAM guidelines, care givers will receive a homebased individualized face to face support provided by breastfeeding peer supporters and phone call support upto 7 weeks post hospital discharge.
  Arms: Breastfeeding peer support intervention.
Other: Standard Care — Caregivers will receive post-discharge support as currently recommended by the World Health Organization (WHO) and national IMAM guidelines.
  Arms: Standard of care

SUMMARY:
The current guidelines used to manage malnutrition among infants aged below 6 months (u6m) recommend that infants admitted to hospital with malnutrition be supported to reestablish exclusive breastfeeding before discharge. Studies have shown that reestablishing exclusive breastfeeding among infants being treated for acute malnutrition is possible. However, follow-up of the infants after discharge has revealed poor growth raising questions about what happens to infant feeding practices after discharge and whether providing breastfeeding support to mothers after discharge would help improve the recovery and growth of their infants.

Providing a package of home-based care with breastfeeding support to mothers of infants u6m recovering from acute malnutrition has the potential to improve the retention of exclusive breastfeeding and lead to enhanced infant growth and survival. To date, no such post-discharge package of care is available in Kenya or other lower and meddle income countries (LMICs). The aim of this study is to apply participatory, qualitative and quantitative approaches to develop and evaluate the impact of a post-discharge package of care on the growth and development of acutely ill malnourished infants after discharge from hospital.

DETAILED DESCRIPTION:
Globally, acute malnutrition affects 8.5 million infants under 6 months of age (u6m). These malnourished infants u6m are at elevated risk of death during admission, death after discharge from hospital and subsequent neurodevelopmental impairment. The 2020 national guidelines for integrated management of acute malnutrition for infants and children (IMAM) recommend that for hospitalised malnourished infants u6m the treatment should focus on re-establishing exclusive breastfeeding (EBF) with discharge when consistent weight gain of >20g/day is achieved on breastmilk alone. In Kilifi, a study to investigate the outcomes of effective guideline implementation, employed breastfeeding peer supporters to facilitate re-establishing exclusive breastfeeding among sick hospitalized malnourished infants u6m.The study achieved 81% infants exclusive breastfeeding by discharge with 67% attaining the World health organization recommended growth velocity on breastmilk alone. However, when infants were followed up 6 weeks after discharge, the criteria for full nutritional recovery, weight adjusted for Length Z score (WFL)>2 were generally not met. Interviews with mothers, breastfeeding peer supporters (BFPS) and health workers at discharge and 4 weeks after discharge suggested that BFPS were central in enabling mothers to achieve exclusive breastfeeding but that mothers found it challenging to maintain exclusive breastfeeding at home after discharge without on-going support. This follow-on study will investigate the hypothesis that providing support during transition from hospital to home environment will help improve nutritional recovery among this vulnerable group of infants. The study will take part in two phases. Phase1 will use participatory and qualitative approaches to develop and pilot test a post-discharge breast-feeding support intervention (BFSI). Phase 2 will involve a randomized control trial to measure the impact of the intervention on growth, EBF and neurodevelopmental outcomes of malnourished infants discharged from hospital following a serious illness.

The primary outcome for the trial is growth (weight gain) assessed at age 6 months, with additional follow up at 9 and 12 months of age to assess mortality, morbidity and neurodevelopmental outcomes. The results of the study will inform efforts to improve post-discharge management of recovering malnourished vulnerable infants u6m.

ELIGIBILITY:
Inclusion Criteria:

Infants admitted to Kilifi County Hospital (KCH) aged between 4 weeks and 12 weeks old

AND Wasting or underweight assessed by Weight-for-length Z-score (WFLz)<-2 OR Weight-for-age Z-score (WFAz) <-2

OR Mid upper arm circumference (MUAC)<110mm OR presence of bilateral pitting oedema AND

* Any possibility to breastfeed (carer of reproductive age willing to breastfeed and infant without clinical abnormalities obstructing breastfeeding
* Caregivers consent to participation in the study

Exclusion Criteria:

Infants with no possibility to breastfeed. OR Infants with congenital abnormalities that would affect breastfeeding e.g. cleft palate or invalidate the use of normal growth standards.

-

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Weight gain | At 26 weeks of age
  The primary outcome for the trial is growth (weight gain) assessed at 26 weeks of age

SECONDARY OUTCOMES:
Morbidity | At 39 weeks and 52 weeks of age
  Assess morbidity at 39 weeks and 52 weeks of age
Mortality | At 39 to 52 weeks of age
  To assess for mortality at the age of 39 to 52 weeks of age

CONTACTS AND LOCATIONS:
Overall Officials: Martha Mwangome, PhD, Principal Investigator — KEMRI WELLCOME TRUST

IPD SHARING:
Plan to Share IPD: Yes
Summary information concerning the study will be posted on the https://clinicaltrials.gov/ platform and on Kenya Medical research Institution (KEMRI)/Wellcome Trust Research Programmes website. Data hosted on the Kemri-Wellcome Trust Research Program (KWTRP) Research Data Repository (https://dataverse.harvard.edu/dataverse/kwtrp will be issued with a Digital Object Identifier (DOI). This can be included as part of a data citation in publications, allowing the datasets underpinning a publication to be identified and accessed. Metadata and documentation about datasets held in KWTRP Data Repository will be publicly searchable and discoverable. Access to the archived data will be managed by the Data Governance committee which receives and reviews requests for both internal and external data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: 3 years
Access Criteria: Apply to the Data Governance Committee: dgc@kemri-wellcome.org

REFERENCES:
- [Background] Kerac M, Blencowe H, Grijalva-Eternod C, McGrath M, Shoham J, Cole TJ, Seal A. Prevalence of wasting among under 6-month-old infants in developing countries and implications of new case definitions using WHO growth standards: a secondary data analysis. Arch Dis Child. 2011 Nov;96(11):1008-13. doi: 10.1136/adc.2010.191882. Epub 2011 Feb 2. PMID 21288999
- [Background] Grijalva-Eternod CS, Kerac M, McGrath M, Wilkinson C, Hirsch JC, Delchevalerie P, Seal AJ. Admission profile and discharge outcomes for infants aged less than 6 months admitted to inpatient therapeutic care in 10 countries. A secondary data analysis. Matern Child Nutr. 2017 Jul;13(3):e12345. doi: 10.1111/mcn.12345. Epub 2016 Jul 25. PMID 27453170
- [Background] Berkley JA, Ngari M, Thitiri J, Mwalekwa L, Timbwa M, Hamid F, Ali R, Shangala J, Mturi N, Jones KD, Alphan H, Mutai B, Bandika V, Hemed T, Awuondo K, Morpeth S, Kariuki S, Fegan G. Daily co-trimoxazole prophylaxis to prevent mortality in children with complicated severe acute malnutrition: a multicentre, double-blind, randomised placebo-controlled trial. Lancet Glob Health. 2016 Jul;4(7):e464-73. doi: 10.1016/S2214-109X(16)30096-1. Epub 2016 Jun 2. PMID 27265353
- [Background] Victora CG, de Onis M, Hallal PC, Blossner M, Shrimpton R. Worldwide timing of growth faltering: revisiting implications for interventions. Pediatrics. 2010 Mar;125(3):e473-80. doi: 10.1542/peds.2009-1519. Epub 2010 Feb 15. PMID 20156903
- [Background] Roberton T, Carter ED, Chou VB, Stegmuller AR, Jackson BD, Tam Y, Sawadogo-Lewis T, Walker N. Early estimates of the indirect effects of the COVID-19 pandemic on maternal and child mortality in low-income and middle-income countries: a modelling study. Lancet Glob Health. 2020 Jul;8(7):e901-e908. doi: 10.1016/S2214-109X(20)30229-1. Epub 2020 May 12. PMID 32405459
- [Background] Vygen SB, Roberfroid D, Captier V, Kolsteren P. Treatment of severe acute malnutrition in infants aged <6 months in Niger. J Pediatr. 2013 Mar;162(3):515-521.e3. doi: 10.1016/j.jpeds.2012.09.008. Epub 2012 Oct 23. PMID 23092531
- [Background] Stewart RC. Maternal depression and infant growth: a review of recent evidence. Matern Child Nutr. 2007 Apr;3(2):94-107. doi: 10.1111/j.1740-8709.2007.00088.x. PMID 17355442
- [Background] Chisti MJ, Graham SM, Duke T, Ahmed T, Faruque AS, Ashraf H, Bardhan PK, Shahid AS, Shahunja KM, Salam MA. Post-discharge mortality in children with severe malnutrition and pneumonia in Bangladesh. PLoS One. 2014 Sep 16;9(9):e107663. doi: 10.1371/journal.pone.0107663. eCollection 2014. PMID 25225798
- [Background] Guideline: Updates on the Management of Severe Acute Malnutrition in Infants and Children. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK190328/ PMID 24649519
- [Background] Health Mo. The Kenya National Intergrated Management of Acute Malnutrition (IMAM) guidelines. 2020
- [Background] McGrath M. Updated review of 46 national guidelines on MAMI: Key findings. London: Emergency Nutrition Network; London School of Hygiene and Tropical Medicine; 2016.
- [Background] Mwangome M, Murunga S, Kahindi J, Gwiyo P, Mwasho G, Talbert A, Kiige L, Samburu B, Mturi N, Abubakar A, Jones C, Berkley JA. Individualized breastfeeding support for acutely ill, malnourished infants under 6 months old. Matern Child Nutr. 2020 Jan;16(1):e12868. doi: 10.1111/mcn.12868. Epub 2019 Aug 2. PMID 31264337
- [Background] Kahindi J, Jones C, Berkley JA, Mwangome M. Establishing exclusive breastfeeding among in-patient malnourished infants in a rural Kenyan hospital: mothers' experiences of a peer supporter intervention. Int Breastfeed J. 2020 May 14;15(1):40. doi: 10.1186/s13006-020-00278-9. PMID 32408904
- [Background] Van Ryneveld M, Mwangome M, Kahindi J, Jones C. Mothers' experiences of exclusive breastfeeding in a postdischarge home setting. Matern Child Nutr. 2020 Oct;16(4):e13016. doi: 10.1111/mcn.13016. Epub 2020 Apr 21. PMID 32319227
- [Background] Chabeda S, Oluoch D, Mwangome M, Jones C. Infant malnutrition treatment in Kenya: Health worker and breastfeeding peer supporter experiences. Matern Child Nutr. 2021 Jul;17(3):e13148. doi: 10.1111/mcn.13148. Epub 2021 Feb 2. PMID 33528108
- [Background] Kenya National Bureau of statistics. Kenya Demographic Health Survey 2014. Kenya National Bureau of Statistics; 2014.
- [Background] Talbert A, Jones C, Mataza C, Berkley JA, Mwangome M. Exclusive breastfeeding in first-time mothers in rural Kenya: a longitudinal observational study of feeding patterns in the first six months of life. Int Breastfeed J. 2020 Mar 5;15(1):17. doi: 10.1186/s13006-020-00260-5. PMID 32138727
- [Background] Eickmann SH, de Lira PI, Lima Mde C, Coutinho SB, Teixeira Mde L, Ashworth A. Breast feeding and mental and motor development at 12 months in a low-income population in northeast Brazil. Paediatr Perinat Epidemiol. 2007 Mar;21(2):129-37. doi: 10.1111/j.1365-3016.2007.00795.x. PMID 17302642
- [Background] O'Sullivan AK, Thompson D, Drummond MF. Collection of health-economic data alongside clinical trials: is there a future for piggyback evaluations? Value Health. 2005 Jan-Feb;8(1):67-79. doi: 10.1111/j.1524-4733.2005.03065.x. PMID 15841896
- [Background] Petrou S. Rationale and methodology for trial-based economic evaluation. . Clinical Investigation. 2012;2(12).
- [Background] Lloyd-Williams H, Edwards RT. Sample size calculation in trials of public health interventions: a discussion of implications for health economists. The Lancet. 2013;382.
- [Background] Harding R, Simms V, Penfold S, McCrone P, Moreland S, Downing J, Powell RA, Mwangi-Powell F, Namisango E, Fayers P, Curtis S, Higginson IJ. Multi-centred mixed-methods PEPFAR HIV care & support public health evaluation: study protocol. BMC Public Health. 2010 Sep 29;10:584. doi: 10.1186/1471-2458-10-584. PMID 20920241
- [Background] Simpson KN, Baran RW, Kirbach SE, Dietz B. Economics of switching to second-line antiretroviral therapy with lopinavir/ritonavir in Africa: estimates based on DART trial results and costs for Uganda and Kenya. Value Health. 2011 Dec;14(8):1048-54. doi: 10.1016/j.jval.2011.06.011. Epub 2011 Nov 6. PMID 22152173
- [Background] Constenla D, Armien B, Arredondo J, Carabali M, Carrasquilla G, Castro R, Durand L, Duran-Arenas L, Garcia ME, Gallegos RV, Gontes ML, Lopez JG, McFarlane C, Montoya R, Sartori AM, Siqueira JB, Martelli CT. Costing Dengue Fever Cases and Outbreaks: Recommendations from a Costing Dengue Working Group in the Americas. Value Health Reg Issues. 2015 Dec;8:80-91. doi: 10.1016/j.vhri.2015.06.001. Epub 2015 Jul 28. PMID 29698176
- [Background] Kirkwood B. R, Sterne JAC. Essential Medical Statistics. Second Edition ed. Oxford: Blackwells publishing Ltd; 2003.
- [Background] Ministry of Health. Guidelines for Prevention of Mother To Child Transmission (PMTCT) of HIV/AIDS in Kenya 2012 [Fourth:[Available from: http://www.faces-kenya.org/wp-content/uploads/2012/11/Guidelines-for-PMTCT-of-HIVAIDS-in-Kenya-1_2012.pdf.
- [Background] WHO, UNICEF. Infant and Young Child Feeding Counselling: An intergrated Course. Geneva: Worls Health Organization; 2006.
- [Background] Corbett M. Severe Malnutrition in the infants less than 6 months: Use of Supplemental Suckling Technique 2000 [Available from: http://fex.ennonline.net/9/tfp.
- [Background] Ministry of Health. National Guidelines for Intergrated Management of Acute Malnutrition 2009 [Available from: http://www.cmamforum.org/Pool/Resources/Kenya-MoH-IMAM-Guideline-June-2009.pdf.
- [Background] Abubakar A, Holding P, van Baar A, Newton CR, van de Vijver FJ. Monitoring psychomotor development in a resource-limited setting: an evaluation of the Kilifi Developmental Inventory. Ann Trop Paediatr. 2008 Sep;28(3):217-26. doi: 10.1179/146532808X335679. PMID 18727851